CLINICAL TRIAL: NCT00760565
Title: A Randomized, Double-Blind, Multiple-Ascending Dose, Placebo-Controlled, Parallel Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO4905417 Following Intravenous Infusion in Healthy Volunteers and Patients With Peripheral Arterial Disease
Brief Title: A Multiple Ascending Dose Study of RO4905417 in Healthy Volunteers and Patients With Peripheral Arterial Disease (PAD).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BP21617
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — inclacumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (12):
- 1 (Experimental)
  Interventions: Drug: RO4905417
- 10 (Placebo Comparator)
  Interventions: Drug: placebo
- 11 (Experimental)
  Interventions: Drug: RO4905417
- 12 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Placebo Comparator)
  Interventions: Drug: placebo
- 3 (Experimental)
  Interventions: Drug: RO4905417
- 4 (Placebo Comparator)
  Interventions: Drug: placebo
- 5 (Experimental)
  Interventions: Drug: RO4905417
- 6 (Placebo Comparator)
  Interventions: Drug: placebo
- 7 (Experimental)
  Interventions: Drug: RO4905417
- 8 (Placebo Comparator)
  Interventions: Drug: placebo
- 9 (Experimental)
  Interventions: Drug: RO4905417

INTERVENTIONS:
Drug: RO4905417 — 3mg/kg iv every 28 days for 3 infusions
  Arms: 1; 3
Drug: RO4905417 — 20mg/kg iv every 28 days for 3 infusions
  Arms: 11; 9
Drug: RO4905417 — 7mg/kg iv every 28 days for 3 infusions
  Arms: 5; 7
Drug: placebo — 3mg/kg iv every 28 days for 3 infusions
  Arms: 2; 4
Drug: placebo — 7mg/kg iv every 28 days for 3 infusions
  Arms: 6; 8
Drug: placebo — 20mg/kg iv every 28 days for 3 infusions
  Arms: 10; 12

SUMMARY:
This single center, multiple ascending dose study will assess the safety, tolerability, pharmacokinetics and pharmacodynamics of RO4905417 at different doses in healthy volunteers and patients with peripheral arterial disease. Three groups of 10 healthy volunteers will receive RO4905417 (either 3mg/kg, 7mg/kg or 20mg/kg) or placebo iv every 28 days for a total of 3 infusions. In addition, two groups of 6 PAD patients will receive RO4905417 (either 3mg/kg, 7mg/kg) or placebo and 1 group of 20 PAD patients will receive 20mg/kg RO4905417 or placebo iv every 28 days for a total of three infusions. The study will have an adaptive design with ongoing assessment of safety and tolerability prior to initiation of the next dose. All subjects will receive 3 doses of RO4905417 or matching placebo at 28 day intervals. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females aged 18-65 years (Arms 1,2,5,6,9,10);
* BMI 18-30kg/m2 (Arms 1,2,5,6,9,10);
* males and females aged 45-75 years with confirmed stable PAD (Arms 3,4,7,8,11,12);
* on a stable dose of statin, aspirin or clopidogrel for at least one month prior to the study (Arms 3,4,7,8,11,12);
* BMI 17.5-35kg/m2 (Arms 3,4,7,8,11,12).

Exclusion Criteria:

* patients with pain at rest and/or local complications;
* history of any cardiovascular event within the previous 6 months;
* treatment with drugs potentially affecting coagulation time or platelet aggregation (except aspirin or clopidogrel);
* evidence of hepatic or renal impairment;
* history of bleeding disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse events; clinical laboratory tests; physical examination; vital signs including ECG. | Throughout study

SECONDARY OUTCOMES:
Pharmacodynamics: bleeding time; protein/vascular markers | Throughout study
Pharmacokinetics of RO4905417 | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (3):
  - Gainesville, Florida
  - Cincinnati, Ohio
  - San Antonio, Texas
- Heidelberg, Australia
- Canada (2):
  - Gatineau, Quebec
  - Montreal, Quebec